CLINICAL TRIAL: NCT02654379
Title: MabThera Drug Utilisation Study and Patient Alert Card Evaluation in Non-Oncology Patients in Europe: An Infusion Centre-Based Approach
Brief Title: Observational Study Evaluating Rituximab Use and Use of the Patient Alert Card in Participants Receiving Rituximab Infusion for a Non-Oncology Indication at Infusion Centers in Europe
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: BA28478
Record Dates: First submitted 2016-01-11; First posted 2016-01-13 (Estimated); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Off-Label Use
MeSH Terms: interventions — Rituximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Cohort: Cohort consisting of participants who are in the center to receive an infusion for rituximab for a non-oncology indication.
  Interventions: Biological: Rituximab

INTERVENTIONS:
Biological: Rituximab — Rituximab use in non-oncology indications
  Other Names: MabThera

SUMMARY:
This study is to characterize the indications for which rituximab is being used and to evaluate the use of the Patient Alert Card (PAC) in participants receiving the medication for non-oncology conditions at infusion centers. The study involves the retrospective chart review of rituximab users' medical records in non-oncology indications as well as a survey to collect information on participant characteristics, and will include questions about participant knowledge on the risk of infections, participant receipt and review of the PAC, and any actions the participant has taken as a result of receiving the PAC.

ELIGIBILITY:
Inclusion Criteria:

* Participant is in the center to receive an infusion for rituximab for a non-oncology indication during the study period
* Aged 18 years or older

Exclusion Criteria:

* Has previously already completed the rituximab survey
* Has participated in the past 12 months in a clinical trial in which rituximab was one of the treatments being evaluated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants in the center to receive an infusion for rituximab for a non-oncology indication during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 1408 (Actual)
Dates: Start 2015-12-18 (Actual); Primary Completion 2017-09-29 (Actual); Study Completion 2017-09-29 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Aware of Known and Potential Risks of Infection Associated with Rituximab | Up to 10 months
Percentage of Participants Using Rituximab Off-Label | Up to 10 months

SECONDARY OUTCOMES:
Disease Activity Score Based on 28 Joints (DAS28) for Participants with Rheumatoid Arthritis (RA) | Up to 10 months
Percentage of Participants Who Received the Patient Alert Card (PAC) | Up to 10 months
Percentage of Participants Who Read the PAC | Up to 10 months
Percentage of Participants Who Received Additional Safety-Related Materials | Up to 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (48):
- France (10):
  - Chu De Clermont Ferrand; Hopital Gabriel Montpied, Clermont-Ferrand
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - Centre Hospitalier Le Mans, Le Mans
  - Hopital Claude Huriez - CHU Lille, Lille
  - Hôpital Lapeyronie, Montpellier
  - CHU NANTES - Hôtel Dieu; Pharmacy, Nantes
  - Hôpital Cochin, Paris
  - Groupe Hospitalier Sud - Hôpital Haut-Lévêque - Centre François Magendie, Pessac
  - CHU Saint-Etienne, Hopital Bellevue, Saint-Etienne
  - CHU de Toulouse - Hôpital Purpan, Toulouse
- Germany (9):
  - Krankenhaus Dresden-Friedrichstadt, Dresden
  - CIRI - Centrum für Innovative Diagnostik und Therapie GmbH, Frankfurt
  - Universitaetsklinikum Freiburg; Innere Medizin II, Gastroenterologie, Freiburg im Breisgau
  - Private Practice Dr. A. Liebhaber, Halle
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Schleswig-Holstein; Campus Lübeck, Lübeck
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz, Mainz
  - Rheumazentrum Ratingen - Studienambulanz, Ratingen
  - Fachkrankenhaus Vogelsang, Vogelsang-Gommern
- Italy (9):
  - Azienda Ospedaliera Universitaria Arcispedale S. Anna, Ferrara, Emilia-Romagna
  - IDI-Istituto Dermopatico dell'Immacolata IRCCS, Rome, Lazio
  - Asst Centro Specialistico Ortopedico Traumato-Logico Gaetano Pini/Cto, Milan, Lombardy
  - Ospedale San Raffaele, Milan, Lombardy
  - Ospedale San Giovanni Bosco, Turin, Piedmont
  - Azienda Ospedaliera Giuseppe Brotzu, Cagliari, Sardinia
  - Azienda Ospedaliera Universitaria Careggi, Florence, Tuscany
  - Azienda Ospedaliero Universitaria Pisana, Pisa, Tuscany
  - A.O.U. Senese Policlinico Santa Maria Alle Scotte, Siena, Tuscany
- Spain (11):
  - Corporacio Sanitaria Parc Tauli, Sabadell, Barcelona
  - Complejo Hospitalario Universitario A Coruña, A Coruña, LA Coruña
  - Hospital Regional Universitario de Malaga; Servicio de Reumatologia, Málaga, Malaga
  - Hospital Meixoeiro, Vigo, Pontevedra
  - Hospital Universitario Virgen Macarena, Seville, Sevilla
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari de Bellvitge; Servicio de Reumatologia, Barcelona
  - Hospital Universitario San Cecilio, Granada
  - Hospital Universitario Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clinico Universitario Valladolid, Valladolid
- United Kingdom (9):
  - Bristol Royal Infirmary, Bristol
  - Addenbrooke's Hospital, Cambridge
  - Southend University Hospital, Colchester
  - Royal Devon and Exeter Hospital (Wonford), Exeter
  - Derriford Hospital, Plymouth
  - Salford Royal, Salford
  - Torbay Hospital, Torquay
  - Royal Cornwall Hospital, Truro
  - New Cross Hospital, Wolverhampton

REFERENCES:
- [Derived] Sarsour K, Beckley-Kartey S, Melega S, Odueyungbo A, Kirchner P, Khalife N, Bangs J. Rituximab utilization for approved and off-label nononcology indications and patients' experiences with the Patient Alert Card. Pharmacol Res Perspect. 2020 Jan 3;8(1):e00555. doi: 10.1002/prp2.555. eCollection 2020 Feb. PMID 31911839